CLINICAL TRIAL: NCT01084031
Title: Dose Titration of Propofol for Tracheal Intubation in Children With Sevoflurane Inhalation Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2009-0470
Record Dates: First submitted 2010-03-05; First posted 2010-03-10 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pediatric Urinary Disorders
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- propofol (Experimental)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — intravenous propofol with sevoflurane inhalation induction

SUMMARY:
Dose titration of propofol for tracheal intubation in children with sevoflurane inhalation induction.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for elective day case surgery were enrolled.

Exclusion Criteria:

* History of obstructive sleep apnea
* Evidence of cardiorespiratory disease
* Those who were obese or allergic to any of the anesthetic agents in this study
* Those with an anticipated difficult airway, full stomach
* History of malignant hyperthermia or other myopathy were excluded.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Assessment of intubation conditions | 30 minutes after the surgery
  Assessment of intubation conditions (vocal cord, intubation condition, cough, movement) , peri-induction HR and BP change, post-operative agitation socre at recovery room. ED50 and ED 95 of each group by uring Dixon's up and down methods.
  peri -induction period -comparison of above factors among each groups (GroupA: ETSevo 3vol%, Group B: ETSevo 3.5vol%, Group: ET Sevo 4vol%)

CONTACTS AND LOCATIONS:
Overall Officials: Hae Keum Kil, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea